CLINICAL TRIAL: NCT04735627
Title: Real-Time Levodopa Monitoring for Improved Management of Parkinson Disease
Brief Title: Real-Time Levodopa Level Monitoring in Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Irene Litvan, Director of the UCSD Parkinson and Other Movement Disorders Center, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201535
Record Dates: First submitted 2020-09-19; First posted 2021-02-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will receive oral carbidopa and levodopa and the minimally invasive experimental device will measure levodopa levels in capillary blood, sweat, and/or interstitial fluid (separate experiments and consents), which will be compared to plasma levodopa levels measured using high-performance liquid chromotography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Levodopameter (Experimental): During the single study visit, participants will receive either: 1) one doses of oral carbidopa/ levodopa. The Levodopameter sensor device will serially measure levodopa levels from either capillary blood, sweat, or interstitial fluid and blood will be simultaneously collected from an intravenous line for high-performance liquid chromotography analysis of plasma levodopa levels.
  Interventions: Device: Levodopameter

INTERVENTIONS:
Device: Levodopameter — There are several minimally-invasive sensors being developed that can detect levodopa levels in the capillary blood, sweat, and interstitial fluid.

SUMMARY:
This project aims to develop a minimally invasive sensor device to monitor levodopa levels in real time. We will test the accuracy, tolerability, and safety of this device in people with Parkinson disease.

DETAILED DESCRIPTION:
People with Parkinson disease (PD) lack the chemical dopamine, which is important for movement. Levodopa replaces dopamine and restores normal motor function in PD. Early in the disease stages, people with PD benefit significantly from levodopa. However, as PD progresses, the brain loses more dopamine-producing cells, which causes motor complications and unpredictable responses to levodopa. To maintain control of symptoms over time, levodopa doses must be increased and given at increasingly shorter intervals. The optimal levodopa regimen is different for each person and may vary from day-to-day, depending on a variety of internal and external factors including meal consumption, activity level, and other lifestyle variances. Currently, clinicians assess levodopa's benefit by the patient's testimony and by clinical exam. However, these methods may not adequately represent the severity or range of complications experienced by the PD patient. Thus, it can be difficult to determine the optimal levodopa treatment regimen, which can cause suboptimal disease management and side effects.

This project aims to develop a continuous, minimally invasive sensor (the "Levodopameter") designed to measure levodopa levels in real time from body fluids (capillary blood, sweat, and interstitial fluid), with the future goals of identifying an individualized treatment regimen for people with PD to improve disease management.

We will compare levodopa levels measured by the Levodopameter to the impractical and expensive "gold standard" high-performance liquid chromatography (HPLC) analysis of plasma levodopa levels. We will first test the device after administering oral carbidopa/levodopa in 10 participants with PD. After that portion of the study is completed and safety confirmed, we will test the device in 10 participants with PD after administering carbidopa and intravenous levodopa. We will also evaluate the device's safety and tolerability.

The long-term goal of this device is to allow PD patients to take proactive measures to assess and maintain an optimal, personalized levodopa regimen, similar to diabetes care in which diabetic patients periodically self-monitor their glucose and adjust their insulin regimen accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must meet the Movement Disorders Society (MDS) diagnostic criteria for clinically established Parkinson disease.
2. Able to provide signed informed consent (in English or Spanish)
3. Mild, moderate, or severe Parkinson disease, able to ambulate (Hoehn and Yahr stages I-IV)
4. Taking instant release oral carbidopa/levodopa therapy
5. Either not taking, or on stable doses of any of the following antiparkinsonian medications: dopamine agonists, monoamine oxidase B (MAO-B) inhibitors or catecholamine O-methyl transferase (COMT) inhibitors

Exclusion Criteria:

1. Other neurological conditions including but not limited to stroke, dementia (including Parkinson disease dementia), or traumatic brain injury
2. Co-existent major psychiatric disease
3. Uncontrolled, active medical conditions (e.g., heart, kidney, or liver failure, diabetes, etc.)
4. Status post deep brain stimulation (DBS) device placement
5. Any other condition, that in the opinion of the investigators, would place the participant at risk.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Levodopa Levels | through study completion, an average of 12 months
  Data analysis from this first-of-its-kind microneedle levodopa monitoring device is necessarily exploratory and descriptive. We will assess the Levodopameter's feasibility and accuracy by comparing its interstitial fluid levodopa measurements to plasma levodopa levels analyzed by high-performance liquid chromatography.

SECONDARY OUTCOMES:
Patient Acceptability of Levodopameter | through study completion, an average of 12 months
  Participants will rate acceptability of the Levodopameter using a symmetric Likert-style questionnaire ranging from 1 (strongly disagree) to 5 (strongly agree) to rate the device's comfort, ease of wear, and other qualities. Averaged acceptability ratings of 4 and higher (agree or strongly agree) would indicate the participant's agreement on the device acceptability.
Device Safety | through study completion, an average of 12 months
  The investigators will monitor for and categorize the adverse events related to the device using the will be classified using the current version of the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Litvan, MD, Principal Investigator — UCSD
Locations (1):
- University of California San DIego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goud KY, Moonla C, Mishra RK, Yu C, Narayan R, Litvan I, Wang J. Wearable Electrochemical Microneedle Sensor for Continuous Monitoring of Levodopa: Toward Parkinson Management. ACS Sens. 2019 Aug 23;4(8):2196-2204. doi: 10.1021/acssensors.9b01127. Epub 2019 Aug 12. PMID 31403773
- [Background] Brunetti B, Valdés-Ramírez G, Litvan I, Wang J. A disposable electrochemical biosensor for L-DOPA determination in undiluted human serum. Electrochemistry Communications 2014. p. 28-31.
- [Background] Bandodkar AJ, Wang J. Non-invasive wearable electrochemical sensors: a review. Trends Biotechnol. 2014 Jul;32(7):363-71. doi: 10.1016/j.tibtech.2014.04.005. Epub 2014 May 19. PMID 24853270
- [Background] Windmiller JR, Wang J. Wearable electrochemical sensors and biosensors: a review.: Electroanalysis; 2013. p. 29-46.

DOCUMENTS (1):
  • Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04735627/ICF_001.pdf